CLINICAL TRIAL: NCT01151384
Title: A Phase 1 Study of Liposome Encapsulated Docetaxel (LE-DT) in Patients With Advanced Solid Tumors
Brief Title: Liposome Encapsulated Docetaxel (LE-DT) in Patients With Solid Tumors
Acronym: LE-DT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: INSYS Therapeutics Inc (Industry)
Responsible Party: Dr. Aquilur Rahman; President & Chief Executive Officer (CEO)., NeoPharm Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LE-DT-101
Record Dates: First submitted 2010-06-23; First posted 2010-06-28 (Estimated); Last update posted 2011-07-04 (Estimated); Status verified 2011-06

CONDITIONS: Solid Tumors
Keywords: Cancer Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LE-DT (Experimental)
  Interventions: Drug: LE-DT

INTERVENTIONS:
Drug: LE-DT — Intravenous infusion, Upto 5 dose levels have been studied i.e. 50, 65, 85, 110 and 132 mg/m2, Every 3 weeks
  Other Names: Liposome Entrapped Docetaxel

SUMMARY:
Liposome Encapsulated Docetaxel (LE-DT) is a novel proprietary delivery system of docetaxel developed by NeoPharm, Inc. In this Phase I study, the LE-DT was evaluated for the maximum tolerated dose and dose limiting toxicity (DLT) in patients with advance solid tumors. It was also evaluated for pharmacokinetic and anti-tumor effects.

DETAILED DESCRIPTION:
Liposome Entrapped Doxetaxel (LE-DT) is a novel, proprietary delivery system of docetaxel developed by NeoPharm, Inc. Docetaxel (currently marketed as Taxotere®) is an anti-microtubule agent that prevents cell division by promoting the assembly and stabilization of microtubules and is used for the treatment of malignancies from breast, prostate, lung, gastric, head and neck. By removing toxic detergent used in Taxotere®, LE-DT showed reduced toxicity and comparable therapeutic efficacy in preclinical studies. In clinic, it is believed that LE-DT will offer advantages to the patient of fewer side effects at similar doses, and possibly greater effectiveness when used at higher doses. In addition, routine premedication to prevent hypersensitivity may not be required.

This study is designed to determine the following:

* The maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of LE-DT.
* The pharmacokinetics of docetaxel following intravenous administration of LE-DT.
* Any anti-tumor effects of LE-DT.

Up to 5 dose levels have been studied.

ELIGIBILITY:
Inclusion Criteria:

* To be included in this study, patients must meet the following criteria:
* Be ≥18 years of age.
* Have advanced (local and/or metastatic) histologically documented cancer considered unresponsive to available conventional modalities or treatments.
* Have an ECOG Performance Status of 0-2.
* Have recovered from acute toxicities of prior treatment:

  * 4 weeks must have elapsed since receiving any investigational agent.
  * 4 weeks must have elapsed since receiving any radiotherapy, or treatment with cytotoxic or biologic agents (≥6 weeks for mitomycin or nitrosoureas). Chronic treatment with non-investigational gonadotropin-releasing hormone analogs or other hormonal or supportive care is permitted.
* >6 months must have elapsed since receiving a high-dose chemotherapy regimen with stem cell support.

  * 2 weeks must have elapsed since any prior surgery or granulocyte-stimulating growth factor therapy.
  * 12 months must have elapsed since any prior treatment with docetaxel. 5. Be in adequate condition as evidenced by the following clinical laboratory values:

    * Absolute neutrophil count (ANC) ≥1,500/mm3.
    * Platelets ≥100,000/mm3.
    * Hemoglobin ≥9.0 g/dL.
    * Albumin ≥3.0 g/dL.
    * Serum creatinine ≤2.0 mg/dL.
    * Total bilirubin ≤1.5 x institutional upper limit normal (ULN).
    * Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase ≤2.5 x ULN.

      6. Patients (male and female) must be willing to practice an effective method of birth control during the study.

      7. Patient or legal representative must understand the investigational nature of this study and sign an Institutional Review Board (IRB)/Independent Ethics Committee approved written informed consent form prior to treatment.

Exclusion Criteria:

* Patients are excluded from this study for the following:

  1. Active uncontrolled bleeding or bleeding diathesis (e.g., active peptic ulcer disease).
  2. Any active infection requiring parenteral or oral antibiotic treatment.
  3. Known infection with human immunodeficiency virus or hepatitis virus.
  4. Active heart disease including myocardial infarction or congestive heart failure within the previous 6 months, symptomatic coronary artery disease, or arrhythmias currently requiring medication.
  5. Known or suspected active central nervous system metastasis. (Patients stable 8 weeks after completion of treatment for central nervous system metastasis are eligible.)
  6. Impending or symptomatic spinal cord compression or carcinomatous meningitis.
  7. Having pre-existing clinically significant neuropathy (NCI CTCAE Grade ≥ 2 neuromotor or Grade ≥ 2 neurosensory) except for abnormalities due to cancer.
  8. Having failed a docetaxel-containing regimen.
  9. Having known non-controllable hypersensitivity to docetaxel or liposomes.
  10. Currently receiving any other standard or investigational treatment for cancer or any other investigational agent for any indication.
  11. Requiring immediate palliative treatment of any kind including surgery and/or radiotherapy.
  12. Female patients who are pregnant or breast-feeding.
  13. Unwilling or unable to follow protocol requirements.
  14. Any condition which, in the Investigator's opinion, deems the patient an unsuitable candidate to receive study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the tolerability and safety | 1 year
  This Phase I, open-label, dose-escalation study was designed to determine the maximum tolerated dose (MTD) of LE-DT in patients with advanced cancer. LE-DT was administered by intravenous infusion, over 1 hour, once every 21 days until occurrence of disease progression or toxicity requiring early treatment discontinuation. Dose escalation was not done until the safety and tolerability at a given dose level has been confirmed.

SECONDARY OUTCOMES:
To evaluate the pharmacokinetic and anti-tumor effect | 1 year
  The patients were evaluated for pharmacokinetic profile upto 48 hours post treatment after cycle 1. The anti-tumor effects were evaluated after every two cycles of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: John L Marshall, MD, Principal Investigator — Georgetowm University Medical Center
Locations (2):
- United States (2):
  - TGEN/Scottsdale Clinical Research Institute, Scottsdale, Arizona
  - Lombardi Comprehensive Cancer Center, Georgetown University, Washington D.C., District of Columbia

REFERENCES:
- [Derived] Deeken JF, Slack R, Weiss GJ, Ramanathan RK, Pishvaian MJ, Hwang J, Lewandowski K, Subramaniam D, He AR, Cotarla I, Rahman A, Marshall JL. A phase I study of liposomal-encapsulated docetaxel (LE-DT) in patients with advanced solid tumor malignancies. Cancer Chemother Pharmacol. 2013 Mar;71(3):627-33. doi: 10.1007/s00280-012-2048-y. Epub 2012 Dec 30. PMID 23274395